CLINICAL TRIAL: NCT04194801
Title: A Muti-center, Open-label, Multiple-dose Phase Ib/II Study to Assess the Safety, Tolerability, Pharmacokinetics, Anti-tumor Efficacy of Fisogatinib(BLU-554) in Combination With CS1001 in Subjects With Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: A Phase Ib/II Study of Fisogatinib(BLU-554) in Subjects With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Collaborators: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS3008-101
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — fisogatinib; sugemalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase Ib: Fisogatinib (BLU-554) 400mg in combination with Sugemalimab (CS1001) 1200mg (Experimental)
  Interventions: Drug: Phase Ib: Fisogatinib (BLU-554) 400mg in combination with Sugemalimab (CS1001) 1200mg
- Phase Ib: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg (Experimental)
  Interventions: Drug: Phase Ib: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg
- Phase II: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg (Experimental)
  Interventions: Drug: Phase II: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg

INTERVENTIONS:
Drug: Phase Ib: Fisogatinib (BLU-554) 400mg in combination with Sugemalimab (CS1001) 1200mg — Phase Ib: participants received 400 mg Fisogatinib (BLU-554) once daily (QD), in combination with 1200mg fixed dose Sugemalimab (CS1001) once every 3 weeks (Q3W). Every 21 days (3 weeks) will be considered as one cycle.
  Arms: Phase Ib: Fisogatinib (BLU-554) 400mg in combination with Sugemalimab (CS1001) 1200mg
Drug: Phase Ib: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg — Phase Ib: participants received 600 mg Fisogatinib (BLU-554) QD, in combination with 1200mg fixed dose Sugemalimab (CS1001) Q3W. Every 21 days (3 weeks) will be considered as one cycle.
  Arms: Phase Ib: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg
Drug: Phase II: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg — Phase II: participants received 600 mg Fisogatinib (BLU-554) QD, in combination with 1200mg fixed dose Sugemalimab (CS1001) Q3W. Every 21 days (3 weeks) will be considered as one cycle.
  Arms: Phase II: Fisogatinib (BLU-554) 600mg in combination with Sugemalimab (CS1001) 1200mg

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetic and efficacy of fisogatinib (formerly known as BLU-554) in combination with CS1001 in patients with locally advanced or metastatic hepatocellular carcinoma (HCC)

ELIGIBILITY:
Inclusion criteria:

1. Voluntarily participate in the clinical study. Fully understand and get informed of this study and sign the Informed Consent Form (ICF).
2. ≥18 years of age on day of signing the informed consent.
3. Unresectable locally advanced or metastatic hepatocellular carcinoma as confirmed by histology or cytology.
4. Stage B or C based on Barcelona Clinic Liver Cancer (BCLC) staging system; In case of Stage B, subject must be ineligible for surgery and/or local therapy, or has progressed after surgery and/or local therapy or refuses surgery and/or local treatment.
5. For Phase Ib, subject has failed after or is unsuitable for the standard systemic therapy against HCC. For Phase II, subject has not previously received systemic therapy.
6. At least one measurable lesion as evaluable by RECIST version 1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1 point.
8. A-level Child-Pugh score.
9. Expected survival≥3 months.
10. For Phase Ib and II, fresh or archived tumor tissue should be provided for analysis in the central laboratory.
11. The function of the main organs was basically normal and met the requirements of the protocol.
12. For subject with HCV infection, HCV antiviral treatment with the locally approved and available HCV antiviral therapy can be received.
13. For subjects with HBV infection, HBV DNA ≤ 2,000 IU/ml at Screening.
14. For female subjects of childbearing potential, serum pregnancy test must be negative within 7 days prior to randomization. Except for female subjects who have been recorded as surgically sterilized or who are postmenopausal, female subjects of childbearing potential or male subjects and their partners must agree to use effective contraception from the signature of the informed consent form (ICF) until at least 6 months after the last dose of study drug.

Exclusion criteria:

1. tumor thrombus in the main portal vein (VP4) by imaging, involving the inferior vena cava or the heart.
2. Prior history of hepatic encephalopathy.
3. History of liver surgery and/or local treatment for HCC (intervention, ablation therapy, absolute alcohol injection, etc.) or radiotherapy, etc. within 4 weeks prior to first dose.
4. Active or documented gastrointestinal bleeding within 6 months (e.g. esophageal or gastric varices, ulcer bleeding).
5. Presence of ascites detected by physical examination or clinical symptoms caused by ascites during the screening period, or ascites that need for special treatment, such as repeated drainage, intraperitoneal drug infusion, etc.
6. Presence of meningeal metastasis or central nervous system (CNS) metastatic lesions.
7. Subject has clinically significant, uncontrolled cardiovascular disease.
8. History of definite interstitial lung disease or non-infectious pneumonia except that caused by local radiotherapy; history of active tuberculosis.
9. Any serious acute, chronic infections that require systemic antimicrobial, antifungal or antiviral therapy at screening, excluding viral hepatitis.
10. Malabsorption syndrome or inability to take the study drug orally for other reasons.
11. Had primary malignancies other than HCC within 5 years.
12. Subject has had major surgery within 4 weeks prior to first dose (procedures such as central venous cannulation, biopsy, and feeding tube placement are not considered as major surgery).
13. Previously received FGFR4 inhibitor treatment.
14. Blood transfusion, use of hematopoietic stimulating factors [including G-CSF (granulocyte colony stimulating factor), GM-CSF (granulocyte-macrophage colony stimulating factor), EPO (erythropoietin) and TPO (thrombopoietin)] and human albumin preparations within 14 days prior to first dose.
15. Requiring corticosteroids (dose equivalent to > 10 mg/day of Prednisone) or other immunosuppressive drugs within 14 days prior to first dose for systemic therapy.
16. Use of traditional Chinese medicine with anti-liver cancer indication within 14 days prior to the first dose.
17. Subject has received potent CYP3A4 inhibitors and/or inducers within 2 weeks prior to first dose.
18. Concurrent HBV and HCV infection.
19. Subjects with known human immunodeficiency virus (HIV) infection.
20. Lactating women.
21. Subjects with a history of hypersensitivity or hypersensitivity to any of the components of the investigational drug.
22. Circumstances that in the opinion of the investigator would preclude participation in the study.
23. Subjects who are unwilling or unable to follow the study procedures as defined.
24. With the exception of alopecia, all toxicities from prior anticancer therapies and other therapies did not recover to ≤ Grade 1 (per CTCAE v5.0) prior to the first dose of study drug.
25. Subjects who have received prior allogeneic stem cell or solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Nanfang Hospital,, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened across 19 centers and enrolled across 11 centers in China. The study consists of 2 parts, including Phase Ib dose escalation and Phase II dose expansion. A total of 26 participants were enrolled in the study and all received ≥ 1 dose of study drug.
Period: Part Ib/II End Of Treatment-BLU554
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Started | 4 | 7 | 15
Completed | 0 | 0 | 0
Not Completed | 4 | 7 | 15
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Radiographic disease progression | 3 | 4 | 9
Not completed — Symptomatic deterioration without radiographic evidence | 0 | 1 | 0
Not completed — Other | 0 | 0 | 2
Not completed — Ongoing treatment | 0 | 0 | 2
Period: Part Ib/II End Of Treatment-CS1001
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Started | 4 | 7 | 15
Completed | 0 | 0 | 0
Not Completed | 4 | 7 | 15
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Radiographic disease progression | 3 | 6 | 9
Not completed — Symptomatic deterioration without radiographic evidence | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1
Not completed — Ongoing treatment | 0 | 0 | 2
Period: Part Ib/II End of Study
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Started | 4 | 7 | 15
Completed | 0 | 0 | 0
Not Completed | 4 | 7 | 15
Not completed — Death | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Study ended by sponsor | 1 | 3 | 8
Not completed — Ongoing treatment | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population consists of all participants receiving at least one dose of investigational product
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Total
Number analyzed (Participants) | 4 | 7 | 15 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 13 | 23
  >=65 years | 0 | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (4.80) | 48.4 (11.82) | 51.6 (12.37) | 49.5 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 3 | 5 | 14 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 7 | 15 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 4 | 7 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Patients With Event(s) of Dose-limiting Toxicity
Description: Number of DLT (Dose-limiting toxicity) During the Administration of BLU-554 in Combination with CS1001. All toxicity or adverse events (AEs) are graded according to NCI-CTCAE 5.0. Any AE occurring during C1 (21 days) that is not clearly caused by something other than investigational drug.
Time Frame: Cycle 1 (21 days) of treatment
Population: Fisogatinib (BLU-554) 600mg arm, 7 subjects were enrolled, of whom 6 completed DLT evaluation and 1 was unevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 6
Participants | 0 | 0

2. Primary Outcome: Phase Ib: Safety and Tolerance
Description: An AE was any untoward medical occurrence after clinical study subjects receive study drug. An SAE was any event that meets any the following criteria: death, life-threatening; inpatient hospitalization or prolongation, persistent or significant disability/incapacity;congenital malformation/birth defects and significant medical events. AE and SAE were graded by CTCAE version 5.0 by severity, from Grade 1 mild to Grade 5 death related AE.
Time Frame: Safety and tolerance assessments continued for the duration of treatment. AEs and SAEs will be collected from time of signature of main informed consent, throughout the treatment period and including the follow-up period, up to approximate 22 months.
Population: Baseline Analysis Population consists of all participants receiving at least one dose of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 7
Participants
  Treatment-Emergent Adverse Event（TEAE） | 4 | 7
  TEAE at least one related to CS1001 or BLU-554 | 4 | 6
  Grade 3-5 TEAE | 2 | 6
  Grade 3-5 TEAE at least one related to CS1001 or BLU-554 | 1 | 4
  Serious TEAE | 1 | 2
  Serious TEAE at least one related to CS1001 or BLU-554 | 0 | 1
  Immune-related TEAE | 2 | 2
  Infusion-related reaction TEAE | 0 | 0
  TEAE Leading to CS1001 rate of infusion modification | 0 | 0
  TEAE Leading to CS1001 dose interruption | 0 | 2
  TEAE Leading to CS1001 permanently discontinuation | 1 | 0
  TEAE Leading to BLU-554 dose reduction | 0 | 2
  TEAE Leading to BLU-554 dose interruption | 1 | 1
  TEAE Leading to BLU-554 permanently discontinuation | 0 | 2
  TEAE Leading to death | 0 | 1

3. Primary Outcome: Phase II: Objective Response Rate (ORR) Assessed by Investigator Based on RECIST Version 1.1
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1 .1) for target lesions and assessed by MRI/ CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), > =30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR. Percentage of subjects who achieve objective tumor response (CR or PR) will be summarized.
Time Frame: Imaging (CT or MRI) assessments per RECIST v1.1 will be performed within 28 days prior to the first dose (baseline assessment), every 9 weeks during the first year of the study, and every 12 weeks thereafter. Up to 22 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 15
Participants
  Responder | 3
  Non-Responder | 12

4. Secondary Outcome: Disease Control Rate Assessed by Investigator
Description: Disease control rate (DCR) is defined as the proportion of participants who achieve complete response (CR), partial response (PR), and stable disease (SD) based on Response Evaluation Criteria In Solid Tumors (RECIST)v1.1. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1 .1) for target lesions and assessed by MRI/ CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), > =30% decrease in the sum of the longest diameter of target lesions. Stable disease(SD) is defined as a tumor that does not meet the criteria for progression or for response.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 7 | 15
Participants | 1 | 3 | 9

5. Secondary Outcome: Duration of Response Assessed by Investigator
Description: Duration of response for responders (CR or PR) is defined as the time interval between the date of the earliest qualifying response and the date of PD or death for any cause (whichever occurs earlier). For subjects who are alive without progression following the qualifying response, duration of response will be censored on the date of last evaluable tumor assessment or last follow-up for progression of disease.
Time Frame: as for outcome 3
Population: Only include participants with confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 0 | 1 | 3
Months |  | 4.34 [NA to NA] — The upper bound and lower bound of the confidence interval could not be calculated | NA [NA to NA] — 1. The median of DOR is not reached 2. The upper bound and lower bound of the confidence interval could not be calculated

6. Secondary Outcome: Phase Ib: Objective Response Rate (ORR) Assessed by Investigator Based on RECIST Version 1.1
Description: as for outcome 3
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Phase Ib: Fisogatinb (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg: Phase Ib: participants received 400 mg Fisogatinib (BLU-554) once daily (QD), in combination with 1200mg fixed dose Sugemalimab (CS1001) once every 3 weeks (Q3W). Every 21 days (3 weeks) will be considered as one cycle.
- Phase Ib: Fisogatinb (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg: Phase Ib: participants received 600 mg Fisogatinib (BLU-554) QD, in combination with 1200mg fixed dose Sugemalimab (CS1001) Q3W. Every 21 days (3 weeks) will be considered as one cycle.
Arm/Group | Phase Ib: Fisogatinb (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinb (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 7
Participants
  Responder | 0 | 1
  Non-Responder | 4 | 6

7. Secondary Outcome: Patients With Anti-CS1001 Antibody
Time Frame: Pre-dose of Cycle 1, 2, 4, 5, 7, 10, 13, 16 and every 8 cycles thereafter. Up to 22 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 7 | 15
Participants | 0 | 0 | 0

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time interval between the date of the first investigational product dose to the date of death from any cause
Time Frame: Subject should be followed from time of registration till the time of subject death. Up to 22 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 7 | 15
Months | 16.2 [8.6 to NA] — The upper bound of the confidence interval could not be estimated because of insufficient number of events. | NA [0.6 to NA] — 1. The median could not be estimated because of insufficient number of events. 2. The upper bound of the confidence interval could not be estimated because of insufficient number of events. | NA [7.1 to NA] — 1. The median could not be estimated because of insufficient number of events. 2. The upper bound of the confidence interval could not be estimated because of insufficient number of events.

9. Secondary Outcome: Disease Control Rate by PD-L1 Protein Level
Time Frame: Imaging (CT or MRI) assessments by FGF19 protein and PD-L1 protein level will be performed within 28 days prior to the first dose (baseline assessment), every 9 weeks during the first year of the study, and every 12 weeks thereafter. Up to 22 months.
Population: Efficacy analysis dataset with dichotomous PD-L1 parameters at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage <1 Percentage; Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage >=1 Percentage; Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage <1 Percentage; Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage >=1 Percentage: Phase II: participants received 600 mg Fisogatinib (BLU-554) QD, in combination with 1200mg fixed dose Sugemalimab (CS1001) Q3W. Every 21 days (3 weeks) will be considered as one cycle.
Arm/Group | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage <1 Percentage | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage >=1 Percentage | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage <1 Percentage | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage >=1 Percentage
Number analyzed (Participants) | 3 | 12 | 14 | 1
Participants | 2 | 7 | 8 | 1

10. Secondary Outcome: Objective Response Rate (ORR) by PD-L1 Protein Level
Time Frame: as for outcome 9
Population: Efficacy analysis dataset with dichotomous PD-L1 parameters at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage <1 Percentage; Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage >=1 Percentage; Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage <1 Percentage; Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage >=1 Percentage: Phase II: patients received 600 mg Fisogatinib (BLU-554) QD, in combination with 1200mg fixed dose Sugemalimab (CS1001) Q3W. Every 21 days (3 weeks) will be considered as one cycle.
Arm/Group | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage <1 Percentage | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With IC Percentage >=1 Percentage | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage <1 Percentage | Phase II: BLU-554 600mg in Combination With CS1001 1200mg With TC Percentage >=1 Percentage
Number analyzed (Participants) | 3 | 12 | 14 | 1
Participants | 1 | 2 | 2 | 1

11. Secondary Outcome: Progression-free Survival Assessed by Investigator
Description: Progression-free Survival is defined as the time from the date of first study dose to disease progression or death (whichever occurs first).
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase II: Fisogatinb (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg: Phase II: participants received 600 mg Fisogatinib (BLU-554) QD, in combination with 1200mg fixed dose Sugemalimab (CS1001) Q3W. Every 21 days (3 weeks) will be considered as one cycle.
Arm/Group | Phase Ib: Fisogatinb (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinb (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinb (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 7 | 15
Months | 2.3 [2.1 to NA] — The upper bound of the confidence interval could not be estimated because of insufficient number of events. | 2.1 [0.6 to 4.1] | 4.1 [1.4 to 6.2]

12. Secondary Outcome: Time to Progression Assessed by Investigator
Description: Time to Progression is defined as the time from the date of first study dose to disease progression. Subjects without event (no disease progression) will be censored at the date of "last tumor assessment".
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase Ib: Fisogatinb (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinb (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinb (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 7 | 15
Months | 2.3 [2.1 to NA] — The upper bound of the confidence interval could not be estimated because of insufficient number of events. | 3.1 [1.1 to NA] — The upper bound of the confidence interval could not be estimated because of insufficient number of events. | 4.2 [1.4 to 6.2]

13. Secondary Outcome: Phase II: Safety and Tolerance
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Baseline Analysis Population consists of all participants receiving at least one dose of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 15
Participants
  Treatment-Emergent Adverse Event（TEAE） | 15
  TEAE at least one related to CS1001 or BLU-554 | 15
  Grade 3-5 TEAE | 7
  Grade 3-5 TEAE at least one related to CS1001 or BLU-554 | 6
  Serious TEAE | 5
  Serious TEAE at least one related to CS1001 or BLU-554 | 3
  Immune-related TEAE | 4
  Infusion-related reaction TEAE | 1
  TEAE Leading to CS1001 rate of infusion modification | 0
  TEAE Leading to CS1001 dose interruption | 6
  TEAE Leading to CS1001 permanently discontinuation | 2
  TEAE Leading to BLU-554 dose reduction | 8
  TEAE Leading to BLU-554 dose interruption | 4
  TEAE Leading to BLU-554 permanently discontinuation | 1
  TEAE Leading to death | 1

14. Secondary Outcome: Pharmacokinetic Parameters of Accumulation Ratio of Fisogatinib (BLU-554)
Description: Pharmacokinetic(PK) parameters of accumulation ratio of Fisogatinib (BLU-554),Rac,AUC. Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For BLU554, Cycle 1 day 1( 0, 0.5 to 24 hour post dose) and Cycle 2 day 1( 0, 0.5 to 24 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg: Participants received 400 mg Fisogatinib (BLU-554) once daily (QD), in combination with 1200mg fixed dose Sugemalimab (CS1001) once every 3 weeks (Q3W). Every 21 days (3 weeks) will be considered as one cycle.
- Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg: Participants received 600 mg Fisogatinib (BLU-554) QD, in combination with 1200mg fixed dose Sugemalimab (CS1001) Q3W. Every 21 days (3 weeks) will be considered as one cycle.
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 5
ratio | 1.22 (36.41) | 1.35 (42)

15. Secondary Outcome: Pharmacokinetic Parameters of Area Under the Serum Concentration-time Curve (AUC) of Fisogatinib (BLU-554)
Description: Pharmacokinetic parameters of area under the serum concentration-time curve (AUC0-τ,ss, Time from 0 to 24h) of Fisogatinib (BLU-554). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For BLU554, Cycle 1 day 1( 0, 0.5 to 24 hour post dose) and Cycle 2 day 1( 0, 0.5 to 24 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*μg/mL
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 11
h*μg/mL | 55.3 (65.43) | 73.8 (29.96)

16. Secondary Outcome: Pharmacokinetic Parameters of Clearance at Steady State (CLss) of Fisogatinib (BLU-554)
Description: Pharmacokinetic Parameters of Clearance at Steady State (Clss) of Fisogatinib (BLU-554). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For BLU554, Cycle 1 day 1( 0, 0.5 to 24 hour post dose) and Cycle 2 day 1( 0, 0.5 to 24 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 11
L/h | 7.24 (65.43) | 8.13 (29.96)

17. Secondary Outcome: Pharmacokinetic Parameters of Maximum Serum Concentration (Cmax) of Fisogatinib (BLU-554)
Description: PK Parameters of Cmax of Fisogatinib (BLU-554). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For BLU554, Cycle 1 day 1( 0, 0.5 to 24 hour post dose) and Cycle 2 day 1( 0, 0.5 to 24 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 15
μg/mL | 7.26 (50.01) | 8.14 (27.52)

18. Secondary Outcome: Pharmacokinetic Parameters of Time to Maximum Serum Concentration (Tmax) of Fisogatinib (BLU-554)
Description: PK Parameters of Tmax of Fisogatinib (BLU-554). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For BLU554, Cycle 1 day 1( 0, 0.5 to 24 hour post dose) and Cycle 2 day 1( 0, 0.5 to 24 hour post dose).
Measure: Median (Full Range); unit: hour
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 4 | 15
hour | 1.53 [0.97 to 3.78] | 2.05 [0 to 3.87]

19. Secondary Outcome: Pharmacokinetic Parameters of Accumulation Ratio of Sugemalimab (CS1001)
Description: PK Parameters of Rac, AUC of Sugemalimab (CS1001). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For CS1001: Cycle 1 day 1(0, 0.5 to 504 hour post dose) and Cycle 4 day 1 (0, 0.5 to 504 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 3 | 2
ratio | 1.1 (67.01) | 2.44 (5.85)

20. Secondary Outcome: Pharmacokinetic Parameters of Area Under the Serum Concentration-time Curve (AUC ) of Sugemalimab (CS1001)
Description: PK Parameters of (AUC 0-τ,ss ) of Sugemalimab (CS1001). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For CS1001: Cycle 1 day 1(0, 0.5 to 504 hour post dose) and Cycle 4 day 1 (0, 0.5 to 504 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*μg/mL
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 1 | 8
h*μg/mL | 148000 (NA) — There is only one person. So, it did not be calculated. | 136000 (34.14)

21. Secondary Outcome: Pharmacokinetic Parameters of Clearance at Steady State (CLss) of Sugemalimab (CS1001)
Description: PK Parameters of CLss of Sugemalimab (CS1001). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For CS1001: Cycle 1 day 1(0, 0.5 to 504 hour post dose) and Cycle 4 day 1 (0, 0.5 to 504 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 1 | 6
L/h | 0.00808 (NA) — There is only one person. So, it did not be calculated. | 0.00821 (23.74)

22. Secondary Outcome: Pharmacokinetic Parameters of Maximum Serum Concentration (Cmax) of Sugemalimab (CS1001)
Description: PK Parameters of Cmax of Sugemalimab (CS1001). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For CS1001: Cycle 1 day 1(0, 0.5 to 504 hour post dose) and Cycle 4 day 1 (0, 0.5 to 504 hour post dose).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 3 | 9
μg/mL | 513 (11.08) | 463 (26.16)

23. Secondary Outcome: Pharmacokinetic Parameters of Time to Maximum Serum Concentration (Tmax) of Sugemalimab (CS1001)
Description: PK Parameters of Tmax of Sugemalimab (CS1001). Only participants with evaluable PK results were included in the analysis. Where data is not presented, the PK profiles were non-measurable. Results for Phase Ib and Phase II have been pooled for the same dosage.
Time Frame: For CS1001: Cycle 1 day 1(0, 0.5 to 504 hour post dose) and Cycle 4 day 1 (0, 0.5 to 504 hour post dose).
Measure: Median (Full Range); unit: hour
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib and Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
Number analyzed (Participants) | 3 | 9
hour | 2.02 [2.0 to 7.3] | 2.12 [1.48 to 7.3]

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data were collected starting at the time of the first dose of study drug, throughout the treatment period and including the safety follow-up period. Up to 22 months.
Arm/Group | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg
All-Cause Mortality (participants affected / at risk) | 2/4 | 3/7 | 3/15
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/7 | 5/15
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg (N=4) | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg (N=7) | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: Fisogatinib (BLU-554) 400mg in Combination With Sugemalimab (CS1001) 1200mg (N=4) | Phase Ib: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg (N=7) | Phase II: Fisogatinib (BLU-554) 600mg in Combination With Sugemalimab (CS1001) 1200mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 5
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 1
Extrasystoles (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Wandering pacemaker (Cardiac disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 12
Nausea (Gastrointestinal disorders) | 1 | 4 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4 | 3
Asthenia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 1 | 6
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Measles (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase decreased (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 3 | 11
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 1
Antinuclear antibody increased (Investigations) | 0 | 1 | 0
Antithrombin III decreased (Investigations) | 0 | 1 | 1
Antithrombin III increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 4 | 10
Bilirubin conjugated increased (Investigations) | 1 | 3 | 7
Bilirubin urine present (Investigations) | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 2 | 1
Blood albumin increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 7
Blood bilirubin increased (Investigations) | 2 | 6 | 12
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 2
Blood cholesterol decreased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 2
Blood fibrinogen increased (Investigations) | 0 | 2 | 1
Blood glucose increased (Investigations) | 1 | 0 | 2
Blood iron increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 1
Fibrin degradation products increased (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 5
Glycocholic acid increased (Investigations) | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Haemoglobin increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 4
Neutrophil count decreased (Investigations) | 1 | 0 | 2
Neutrophil count increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 2 | 0 | 6
Protein urine present (Investigations) | 1 | 2 | 3
Prothrombin time prolonged (Investigations) | 0 | 2 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 1
Red blood cell sedimentation rate decreased (Investigations) | 0 | 1 | 0
Total bile acids increased (Investigations) | 0 | 2 | 1
Tri-iodothyronine free increased (Investigations) | 0 | 1 | 0
Tri-iodothyronine increased (Investigations) | 0 | 1 | 0
Urobilinogen urine increased (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 0 | 3
Weight increased (Investigations) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 1 | 3
White blood cell count increased (Investigations) | 0 | 0 | 1
Copper deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT04194801/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT04194801/SAP_001.pdf